CLINICAL TRIAL: NCT00029172
Title: Treatment for Post-Stroke Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Linda Williams, M.D., Roudebush VA Medical Center
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: 9903-06
Record Dates: First submitted 2002-01-08; First posted 2002-01-09 (Estimated); Results first posted 2010-01-28 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2009-12

CONDITIONS: Stroke; Depression
Keywords: stroke; depression
MeSH Terms: conditions — Stroke; Depression | interventions — Case Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nurse Case management (Experimental)
  Interventions: Other: case management

INTERVENTIONS:
Other: case management

SUMMARY:
The purpose of this study is to evaluate a program of education, medicine, and monitoring for the treatment of depression after a stroke.

DETAILED DESCRIPTION:
This trial will compare outcomes in depressed patients receiving the Activate-Initiate-Monitor (AIM) intervention vs. those receiving usual care, and will also compare outcomes in depressed and non-depressed stroke survivors. Patients are screened for depression 1 to 2 months post-stroke. Patients with depression are then randomized to the AIM intervention or control group. Patients without depression are also enrolled at the same time and are matched by hospital site to the depressed patients.

The AIM intervention is a 3-part program consisting of activating or educating the patient and his/her family about post-stroke depression, instituting treatment for depression, and monitoring antidepressant treatments for side effects, efficacy, and compliance. Control patients are evaluated and treated with usual care by their physicians. Patients without depression do not receive the intervention but complete the same assessments on the same schedule as the patients with depression.

ELIGIBILITY:
* No severe language or cognitive deficits,
* life expectancy of at least 9 months, and
* willingness to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 1999-05; Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Williams, M.D., Principal Investigator — Roudebush VA Medical Center Health Services Research and Development 11H
Locations (4):
- United States (4):
  - Indiana University Hospital, 550 N. University Blvd., Indianapolis, Indiana
  - Methodist Hospital of Indiana, 1601 N. Capitol, Indianapolis, Indiana
  - Roudebush VA Medical Center, Health Services Research and Development 11H, 1481 W. 10th Street, Indianapolis, Indiana
  - Wishard Memorial Hospital, 1001 W. 10th Street, Indianapolis, Indiana

REFERENCES:
- [Background] Williams LS, Brizendine EJ, Plue L, Bakas T, Tu W, Hendrie H, Kroenke K. Performance of the PHQ-9 as a screening tool for depression after stroke. Stroke. 2005 Mar;36(3):635-8. doi: 10.1161/01.STR.0000155688.18207.33. Epub 2005 Jan 27. PMID 15677576
- [Background] Williams LS, Bakas T, Brizendine E, Plue L, Tu W, Hendrie H, Kroenke K. How valid are family proxy assessments of stroke patients' health-related quality of life? Stroke. 2006 Aug;37(8):2081-5. doi: 10.1161/01.STR.0000230583.10311.9f. Epub 2006 Jun 29. PMID 16809575
- [Result] Williams LS, Kroenke K, Bakas T, Plue LD, Brizendine E, Tu W, Hendrie H. Care management of poststroke depression: a randomized, controlled trial. Stroke. 2007 Mar;38(3):998-1003. doi: 10.1161/01.STR.0000257319.14023.61. Epub 2007 Feb 15. PMID 17303771

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 4 Indianapolis based hospitals. Depression enrollment and screening occurred between 1 and 2 months post stroke.
Period: Overall Study
Arm/Group | Case Management
Started | 188
Completed | 182
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Case Management
Number analyzed (Participants) | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99
  Male | 83
Region of Enrollment [Number; unit: participants]
  United States | 182

OUTCOME MEASURES:

1. Primary Outcome: Twelve Week Depression Outcomes
Description: Depression remission was defined as HAM-D less than 8 or HAM-D decreased by 50%.
  The Hamilton Rating Scale for Depression is measured on a scale from no depression - major depression, 0-52 units on a scale.
Time Frame: Twelve week
Measure: Mean (Standard Deviation); unit: HAM-D depression score
Arm/Group | Case Management
Number analyzed (Participants) | 182
HAM-D depression score | 10.6 (6.9)

ADVERSE EVENTS:
Arm/Group | Case Management
Serious Adverse Events (participants affected / at risk) | 0/182
Other Adverse Events (participants affected / at risk) | 0/182

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No